CLINICAL TRIAL: NCT06877676
Title: Pre-Approval Access US Intermediate Size Expanded Access Protocol for TAR-200 Treating Physician Use
Brief Title: Pre-Approval Expanded Access Study for TAR-200 Treating Physician Use
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 17000139BLC4003; 17000139BLC4003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Non-Muscle Invasive Bladder Neoplasms
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: TAR-200 — Participants will undergo insertion of TAR-200 transurethrally into the bladder via catherization using the co-packed urinary placement catheter only in accordance with the Instructions for Use (IFU).

SUMMARY:
The purpose of this pre-approval access program is to provide access to TAR-200 prior to its marketing authorization for the treatment of participant(s) with high-risk non-muscle invasive bladder cancer (HR-NMIBC).

ELIGIBILITY:
Inclusion criteria:

* Participant has exhausted all clinically appropriate alternative forms of treatment and is not eligible for, or does not have access to, a clinical trial
* Histologically confirmed diagnosis of persistent or recurrent high-risk non-muscle-invasive bladder cancer (HR-NMIBC), carcinoma in situ (CIS) (OR Tis) with or without papillary disease (T1, high-grade Ta), within 12 months of completion of the last dose of BCG therapy, in participants who have received adequate Bacillus Calmette-Guérin (BCG)
* All visible papillary disease must be fully resected (absent) prior to initiation of treatment
* Participants must be ineligible for or have elected not to undergo Radical Cystectomy (RC)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status Grade of 0, 1, or 2

Exclusion criteria:

* Presence or history of histologically confirmed, muscle invasive, locally advanced, nonresectable, or metastatic urothelial carcinoma (that is, T2, T3, T4, and/or Stage IV)
* Presence of any bladder or urethral anatomic feature that, in the opinion of the Investigator, may prevent the safe placement, indwelling use, or removal of TAR-200. Participants with tumors involving the prostatic urethra in men will be excluded
* Evidence of bladder perforation during diagnostic cystoscopy
* A history of clinically significant polyuria with recorded 24-hour urine volumes greater than 4000 milliliters (>4000 mL)
* Active malignancies (i.e., progressing or requiring treatment change in the last 24 months) other than HR-NMIBC

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC